CLINICAL TRIAL: NCT06820086
Title: The Pragmatic EE-PRS Trial Assessing Polygenic Risk Driven Statin Therapy for Cardiovascular Disease Prevention
Brief Title: Polygenic Risk Driven Pragmatic Statin Trial for Heart Disease Prevention
Acronym: EE-PRS
Status: Enrolling by invitation | Phase: Phase 4 | Type: Interventional
Sponsor: Mikk JÜRISSON (Other)
Collaborators: Funding: European Union (the sponsor does not fund the study) (Unknown); The Estonian Health Insurance Fund (Unknown); North Estonian Medical Center (Unknown); Tartu University Hospital (Other)
Responsible Party: Sponsor-Investigator, Mikk JÜRISSON, Associate professor of Public Health, University of Tartu
Organization: University of Tartu (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: EEPRS12308; 2024-513424-42-01 (EU CTIS Number)
Record Dates: First submitted 2025-01-22; First posted 2025-02-11 (Actual); Last update posted 2025-03-25 (Actual); Status verified 2025-03

CONDITIONS: PRS-based Primary Prevention of CVD
Keywords: Polygenic Risk Score; Statin Treatment for Primary Prevention; High Polygenic Risk Score for Coronary Artery Disease
MeSH Terms: conditions — Genetic Risk Score | interventions — Rosuvastatin Calcium

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Intervention arm receiving statin treatment (Experimental): Intervention arm participants (n=1250) comprise healthy men aged 45- 80 years and women aged 55-80 years with a high (top 20%) coronary artery disease (CAD) polygenic risk score.
  They are prescribed by their primary care physician the trial medication, rosuvastatin 20mg, 1 tablet per day, for the entire duration of the trial. Intervention arm participants will be measured and regular blood analyses will be taken throughout the trial. They will be having regular primary care visits with their family physician and telemedicine visits with study nurses.
  Interventions: Drug: Rosuvastatin 20mg
- Control arm (No Intervention): Control arm participants (n=1250) comprise healthy men aged 45- 80 years and women aged 55-80 years with a high (top 20%) coronary artery disease (CAD) polygenic risk score.
  Participants in the control arm of the trial will be following regular primary care as their family doctors will not be informed of their patients' participation in the trial. This means that in the control arm real-life primary care activities will take place including potential cholesterol-lowering treatment based on the current treatment and prevention guidelines. At the end of the trial, physicians will be informed about their patients who were in the control arm for scheduling a final study visit and ordering a blood test. During the final trial visit the physicians will inform participants of their CAD PRS, provide counselling and take final measurements.

INTERVENTIONS:
Drug: Rosuvastatin 20mg — Preventive statin treatment with rosuvastatin 20mg, 1 tablet per day, for healthy individuals with top 20% CAD PRS.
  Arms: Intervention arm receiving statin treatment

SUMMARY:
This research investigates the potential advantages of intensive preventive statin treatment for healthy men aged 45-80 and women aged 55-80 who possess a high genetic predisposition to coronary artery disease (CAD). By specifically targeting the top 20% of individuals with elevated CAD polygenic risk scores (PRS), the study seeks to find out whether this tailored approach can notably decrease the occurrence of cardiovascular disease and mortality over a five-year period when compared with usual care. Despite the potential of PRS in pinpointing individuals at heightened risk for cardiovascular disease, there is a lack of focused and prospective investigations in existing research. This study aims to bridge this gap by examining whether preventive statin therapy for individuals with high CAD PRS is not only effective in diminishing cardiovascular events but also economically viable. The comparison between the statin treatment arm and standard care practice is conducted in a pragmatic manner at the primary care level.

ELIGIBILITY:
Inclusion Criteria:

* Men aged 45-80 on 1 January 2025
* Women aged 55-80 on 1 January 2025
* CAD PRS top 20% confirmed by the Estonian Biobank (we intend to sample top 15% PRS individuals but we might have to also include 15-20% PRS individuals to fulfil the required sample size)
* The family physician of the study participant has been contracted to participate in the trial
* Written informed consent has been provided to participate in the trial

Exclusion Criteria:

* Diagnosed with ischemic heart disease (I20-I25), stroke or transient ischemia (I60-64, I69, G45), peripheral vascular occlusion (I65-66, I67.2, I70, I73.9), diseases of liver (K70-K77), end stage renal disease (N18.0), mental and behavioural disorders due to psychoactive substance use (F10-F19).

  -- The diagnosis must be present at least 2 times on a health claim or prescription within at least a 6-month period between 1.01.2022-31.12.2024.
* Currently using statin treatment:

  * The individual has at least 1 prescription from ATC groups C10AA or C10BA between 01.01.2022- 31.12.2024.
  * The individual has answered in the recruitment call that he/she is currently using statins or has been prescribed statins in the past 3 years.
* Has familiar hypercholesterolemia (APOB, PCSK9, LDLR genes verified by the Estonian biobank)
* Is currently participating in other clinical trials.
* Has been taking investigative trial medication during the past 30 days prior to study inclusion.
* Co-morbid physical or mental illnesses that prevent the individual from granting consent or participating in the trial (according to the judgement of the investigator).
* Individuals taking:

  * a combination of sofosbuvir/velpatasvir/voxilaprevir (used to treat hepatitis C);
  * ciclosporin
  * fusidic acid orally or by injection.
* Individuals with a substance abuse disorder (alcohol, narcotic substances).
* Individuals with hypersensitivity to the active substance (rosuvastatin or atorvastatin) or its excipients.

Ages: 45 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2500 (Estimated)
Dates: Start 2025-04 (Estimated); Primary Completion 2030-02 (Estimated); Study Completion 2033-02 (Estimated)

PRIMARY OUTCOMES:
Time to the first occurrence of Major Adverse Cardiovascular Events (MACE). | From enrollment to three years after the end of treatment.
  Time to the first occurrence of Major Adverse Cardiovascular Events (MACE), ICD-10 codes: ischaemic heart disease (I20-I25), stroke or transient ischemia (I60-64, I69, G45), peripheral vascular occlusion (I65-66, I67.2, I70, I73.9), revascularization (Z95.1, Z95.5, Z95.8, Z95.9) or cardiovascular death (I00-78) from baseline.

SECONDARY OUTCOMES:
Incidence rate of death from any cause among the study participants | From enrollment to three years after the end of treatment.
Change in CVD risk factors from baseline by the end of the trial in the intervention and control arm; | From enrollment to the end of treatment at 5 years.
  Change in CVD risk factors from baseline (LDL-cholesterol, blood pressure, BMI, waist circumference, smoking, alcohol consumption prevalence) by the end of the trial in the intervention and control arm;
Treatment adherence in the intervention arm. | From enrollment to the end of treatment at 5 years.
  Treatment adherence in the intervention arm based on prescriptions and purchases of statins (C10AA, C10BA) and self-reporting using the MARS-5 scale
Fidelity of intervention implementation. | From enrollment to the end of treatment at 5 years.
  Intervention fidelity will be calculated as a composite score by combining adherence rates (proportion of prescribed activities completed) and participant feedback (average satisfaction and engagement ratings from online questionnaires).
Acceptability of the primary prevention program across study participants measured using an online questionnaire assessing satisfaction, perceived relevance, and ease of participation. | From first study visit to the end of treatment at 5 years.
Satisfaction with study processes and results measured using an online questionnaire assessing satisfaction, perceived relevance, and ease of participation. | From study enrollment to the end of treatment at 5 years.
Difference in plasma concentrations of rosuvastatin. | From enrollment to month 3 of treatment.
  Difference in plasma concentrations of rosuvastatin comparing study participants with and without a mutation in the SLCO1B1, ABCG2, CYP2C9, CYP2C19, UGT-d, SLCO1B3, SLCO2B1, ABCC2, ABCB11 genes.
Difference in rosuvastatin side effects. | From enrollment to the end of treatment at 5 years.
  Difference in rosuvastatin side effects between study participants with and without a mutation in the SLCO1B1, ABCG2, CYP2C9, CYP2C19, UGT-d, SLCO1B3, SLCO2B1, ABCC2, ABCB11 genes.
Utilisation of healthcare resources evaluated through a cost-utilty model | From enrollment to the end of treatment at 5 years.
  Data on healthcare resource utilization, including non-trial physician and cardiologist visits, hospitalizations, length of stay, informal care, and direct healthcare costs, will be aggregated to develop a cost-utility model.
Number of participants with adverse events and serious adverse events from statin therapy. | From enrollment to the end of treatment at 5 years.
Number of participants who withdrew or dropped out from the study. | From enrollment to the end of treatment at 5 years.
Utilities from the EQ-5L-5D surveys and productivity costs from the iPCQ survey for calculating quality-adjusted life years (QALY) gained over a lifetime, incremental cost-effectiveness ratio (ICER). | From enrollment to the end of treatment at 5 years.

OTHER OUTCOMES:
Association of microbial species, functional diversity, and statin side effect risk, measured by species count and functional diversity. | From enrollment to three years after the end of treatment.
  Microbiome composition and functionality will be profiled using the bioBakery four toolkit. Taxonomic annotation will be carried out using the MetaPhlAn4 software, and functional annotation will be done using the HUMAnN 3.0 software. Microbiome diversity will be assessed using the observed number of microbial species and the Shannon diversity index. Functional diversity will be characterized using the number of unique UniRef90 gene families. Centered log-ratio transformed (CLR) abundances of microbial species and gene families are used for univariate analysis. Species and gene families prevalent in more than 5% of the samples are considered for the study. Half the minimal non-zero relative abundance of species and gene family level dataset are used for zero-imputation before the CLR transformation.

CONTACTS AND LOCATIONS:
Overall Officials: Mikk Jürisson, PhD, Study Director — Institute of Family Medicine and Public Health, University of Tartu; Aet Elken (Saar), PhD, Principal Investigator — Heart Clinic, Tartu University Hospital; Margus Viigimaa, PhD, Principal Investigator — North Estonia Medical Centre
Locations (2):
- Estonia (2):
  - North Estonia Medical Centre, Tallinn, Harju
  - Tartu University Hospital, Tartu, Tartu

IPD SHARING:
Plan to Share IPD: No